CLINICAL TRIAL: NCT00613652
Title: A Phase I, Open-Label, Dose-Escalation Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD4877 Administered Weekly in Japanese Adult Patients With Advanced Solid Malignancies
Brief Title: A Phase I, Dose-Escalation Study to Assess the Safety and Drug Levels in Blood of AZD4877 in Japanese Adult Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D2782C00008
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2009-07-21 (Estimated); Status verified 2009-07

CONDITIONS: Cancer; Tumors; Carcinoma
Keywords: solid tumors; solid malignancies
MeSH Terms: conditions — Neoplasms; Carcinoma | interventions — N-(3-aminopropyl)-N-(1-(5-benzyl-3-methyl-4-oxo-(1,2)thiazolo(5,4-d)pyrimidin-6-yl)-2-methylpropyl)-4-methylbenzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: AZD4877 — 10 mg IV (3 weeks treatment 1 week rest)

SUMMARY:
The primary purpose of this study is to evaluate the safety and tolerability of AZD4877 on a weekly schedule in Japanese patients with advanced solid malignancies

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with solid tumour but which have no standard treatment or did not respond to previous treatments.
* Patients who usually have mild symptoms capable of walking and light and sedentary work.
* Patients who can stay in hospital at least during 4 weeks.

Exclusion Criteria:

* Patients who have received treatment with anti-cancer agent within 4 weeks prior to first dose of study treatment; 6 weeks if the anti-cancer agent is mitomycin.
* Patients with abnormally low levels of neutrophil count, platelet count, or haemoglobin, indicators of bone marrow function.
* Patients who received therapeutic radiotherapy at central nervous system within 3 months prior to first dose of study treatment; the other sites within 4 weeks; or local site within 2 weeks.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of AZD4877 on a weekly schedule in Japanese patients with advanced solid malignancies | weekly

SECONDARY OUTCOMES:
To determine the PK profile of AZD4877 on a weekly schedule in Japanese patients with advanced solid malignancies | weekly

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Fukuoka, Japan